CLINICAL TRIAL: NCT05532904
Title: Evaluation and Comparison of Multidisciplinary Day-hospital Versus Waiting List Management of Persistent Symptoms After an Acute Episode of COVID-19
Brief Title: Multidisciplinary Day-hospital Versus Waiting List Management of Post-COVID-19 Persistent Symptoms (ECHAP-COVID)
Acronym: ECHAP-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP220357; 2022-A00268-35 (Other: ID-RCB Number)
Record Dates: First submitted 2022-07-12; First posted 2022-09-08 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Post COVID-19 Condition
Keywords: Randomized controlled trial; Cognitive behavior therapy; Physical exercise; Cognitive remediation; Post covid-19 condition
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): This 6-week program of care will include:
  * group education sessions including a psycho-education component (1 session / week)
  * a personalized exercise training protocol (from 1 session of supervision to 3 sessions of guided exercise per week) adapted to the results of the VO2max exercise test.
  * if dysfunctional health beliefs are identified (SSD-12 score ≥ 26): a group protocol of cognitive and behavior therapy (2 sessions per week, including at least 1 in person).
  * if cognitive complaints and/or neuropsychological impairment: a cognitive remediation protocol (1 group session plus 2 home sessions per week)
  Interventions: Behavioral: Personalized multidisciplinary day-hospital intervention
- Control (No Intervention): Usual care (waiting list)

INTERVENTIONS:
Behavioral: Personalized multidisciplinary day-hospital intervention — This 6-week program of care will include:
  * group education sessions including a psycho-education component (1 session / week)
  * a personalized exercise training protocol (from 1 session of supervision to 3 sessions of guided exercise per week) adapted to the results of the VO2max exercise test.
  * if dysfunctional health beliefs are identified (SSD-12 score ≥ 26): a group protocol of cognitive and behavior therapy (2 sessions per week, including at least 1 in person).
  * if cognitive complaints and/or neuropsychological impairment: a cognitive remediation protocol (1 group session plus 2 home sessions per week)
  Arms: Intervention

SUMMARY:
After an acute episode of COVID-19, many patients experience persistent or recurrent symptoms with substantial impairment of their quality of life. The most common symptoms are fatigue, dyspnea, cognitive impairment and pain, but symptoms of all types have been reported. The heterogeneity of symptoms and their potential pathophysiology makes individualized and multidisciplinary management essential.

The primary objective of this study is to evaluate the change in quality of life at 6 months in patients with persistent symptoms after an acute episode of COVID-19 after 6 weeks of personalized multidisciplinary outpatient management versus usual care.

DETAILED DESCRIPTION:
After an acute episode of COVID-19, many patients experience persistent or recurrent symptoms with substantial impairment of their quality of life. The most common symptoms are fatigue, dyspnea, cognitive impairment, and pain, but symptoms of all types have been reported. The heterogeneity of symptoms and their potential pathophysiology makes individualized and multidisciplinary management essential.

The primary objective is to evaluate the change in quality of life at 6 months in patients with persistent symptoms after an acute episode of COVID-19 after 6 weeks of personalized multidisciplinary outpatient management versus usual care. The secondary objectives are to evaluate the evolution of the quality of life at 3 months, the evolution of the main persistent symptoms (fatigue, dyspnea, cognitive complaints, pain), the patients' satisfaction, the predictive and explanatory factors of the evolution.

This is a prospective randomized open-label study in two parallel arms: personalized multidisciplinary outpatient intervention versus usual care (waiting list). This 6-week program of care will include:

* group education sessions including a psycho-education component (1 session / week)
* a personalized exercise training protocol (from 1 session of supervision to 3 sessions of guided exercise per week) adapted to the results of the VO2max exercise test
* if dysfunctional health beliefs are identified (SSD-12 score ≥ 26): group cognitive and behavior therapy (2 sessions per week, including at least 1 in person).
* if cognitive complaints and/or neuropsychological impairment: a cognitive remediation protocol (1 group session plus 2 home sessions per week)

ELIGIBILITY:
Inclusion Criteria:

* Having had an initial episode of symptomatic COVID-19 according to one of the following criteria:

  * SARS-Cov-2 PCR +
  * SARS-Cov-2 + antigenic test
  * SARS-Cov-2 + serology
  * Prolonged anosmia/ageusia of sudden onset
  * Typical chest CT scan
* Still having at least one of the initial symptoms and possibly new symptoms including fatigue, dyspnea, cognitive impairment or pain beyond 4 weeks after the onset of the acute phase of the disease.
* These initial and persistent symptoms are not better explained by another diagnosis not known to be related to Covid-19.
* These symptoms are the cause of an alteration in quality of life and global functioning deemed significant by the patient.
* Having an indication to either supervised exercise and / or cognitive behavior therapy and / or cognitive remediation Exclusion Criteria
* Medical emergency requiring management not compatible with research
* Neuropsychiatric disorder likely to alter cognitive functions, prior to the Covid-19 episode
* Medical contraindication to exercise training such as pericarditis or progressive myocarditis
* Patient under state medical assistance
* Patient who does not speak French
* Pregnancy in progress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Quality of life | at 6 Months
  SF-12 global score - 12-item Short Form Survey (SF-12) is a general health questionnaire. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12)

SECONDARY OUTCOMES:
Quality of life | at 3 Months
  SF-12 global score - 12-item Short Form Survey (SF-12) is a general health questionnaireTwo summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12)
Fatigue | at 3 months, 6 months
  Pichot's scale global score - may vary between 0 and 32. A score above 22 reveals excessive fatigue
Dyspnea | at 3 months, 6 months
  Borg scale (0 min-10 max)
Cognitive complaint | at 3 months, 6 months
  Mac Nair & Kahn (1983) cognitive difficulties questionnaire, French GRECO consensus version
Pain | at 3 months, 6 months
  Numerical rating scale - from 0 (no pain) to 10 (the maximum imaginable pain)
Patient's satisfaction | at 3 months, 6 months
  Ad hoc questionnaire
Physical fitness | at inclusion, 3 months, 6 months
  Global physical activity questionnaire (GPAQ) score
Post-effort heart rate | at inclusion, 3 months, 6 months
  Difference between estimated and measured heart rate (HR) at the end of the walking test
Weight loss | at inclusion, 3 months, 6 months
  % weight loss
BMI | at inclusion, 3 months, 6 months
  BMI
Blood albumin | at inclusion, 3 months, 6 months
  Blood albumin
Nutritional risk | at inclusion, 3 months, 6 months
  Nutritional risk index
Health beliefs associated with persistent symptoms | at inclusion, 3 months, 6 months
  SSD-12 global score- may vary between 0 and 48 points - Each of the three psychological sub-criteria of DSM-5 somatic symptom disorder (cognitive, affective, behavioral) is measured by four items with all item scores ranging between 0 and 4 (0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = very often) Ratings are summed up to make a simple sum score

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Lemogne, MD, PhD, Principal Investigator — AP-HP and Université Paris Cité
Locations (1):
- Hôtel Dieu Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alonso-Lana S, Marquie M, Ruiz A, Boada M. Cognitive and Neuropsychiatric Manifestations of COVID-19 and Effects on Elderly Individuals With Dementia. Front Aging Neurosci. 2020 Oct 26;12:588872. doi: 10.3389/fnagi.2020.588872. eCollection 2020. PMID 33192483
- [Background] Crook H, Raza S, Nowell J, Young M, Edison P. Long covid-mechanisms, risk factors, and management. BMJ. 2021 Jul 26;374:n1648. doi: 10.1136/bmj.n1648. PMID 34312178
- [Background] Varatharaj A, Thomas N, Ellul MA, Davies NWS, Pollak TA, Tenorio EL, Sultan M, Easton A, Breen G, Zandi M, Coles JP, Manji H, Al-Shahi Salman R, Menon DK, Nicholson TR, Benjamin LA, Carson A, Smith C, Turner MR, Solomon T, Kneen R, Pett SL, Galea I, Thomas RH, Michael BD; CoroNerve Study Group. Neurological and neuropsychiatric complications of COVID-19 in 153 patients: a UK-wide surveillance study. Lancet Psychiatry. 2020 Oct;7(10):875-882. doi: 10.1016/S2215-0366(20)30287-X. Epub 2020 Jun 25. PMID 32593341
- [Background] Gouraud C, Bottemanne H, Lahlou-Laforet K, Blanchard A, Gunther S, Batti SE, Auclin E, Limosin F, Hulot JS, Lebeaux D, Lemogne C. Association Between Psychological Distress, Cognitive Complaints, and Neuropsychological Status After a Severe COVID-19 Episode: A Cross-Sectional Study. Front Psychiatry. 2021 Sep 3;12:725861. doi: 10.3389/fpsyt.2021.725861. eCollection 2021. PMID 34539470
- [Background] Taquet M, Luciano S, Geddes JR, Harrison PJ. Bidirectional associations between COVID-19 and psychiatric disorder: retrospective cohort studies of 62 354 COVID-19 cases in the USA. Lancet Psychiatry. 2021 Feb;8(2):130-140. doi: 10.1016/S2215-0366(20)30462-4. Epub 2020 Nov 9. PMID 33181098
- [Background] Klem F, Wadhwa A, Prokop LJ, Sundt WJ, Farrugia G, Camilleri M, Singh S, Grover M. Prevalence, Risk Factors, and Outcomes of Irritable Bowel Syndrome After Infectious Enteritis: A Systematic Review and Meta-analysis. Gastroenterology. 2017 Apr;152(5):1042-1054.e1. doi: 10.1053/j.gastro.2016.12.039. Epub 2017 Jan 6. PMID 28069350
- [Background] Brascher AK, Schulz SM, Van den Bergh O, Witthoft M. Prospective study of nocebo effects related to symptoms of idiopathic environmental intolerance attributed to electromagnetic fields (IEI-EMF). Environ Res. 2020 Nov;190:110019. doi: 10.1016/j.envres.2020.110019. Epub 2020 Aug 7. PMID 32777274
- [Background] De Peuter S, Van Diest I, Lemaigre V, Li W, Verleden G, Demedts M, Van den Bergh O. Can subjective asthma symptoms be learned? Psychosom Med. 2005 May-Jun;67(3):454-61. doi: 10.1097/01.psy.0000160470.43167.e2. PMID 15911910
- [Background] Graeupner D, Coman A. The dark side of meaning-making: How social exclusion leads to superstitious thinking. Journal of Experimental Social Psychology. 1 mars 2017;69:218-22.
- [Background] Madden VJ, Harvie DS, Parker R, Jensen KB, Vlaeyen JW, Moseley GL, Stanton TR. Can Pain or Hyperalgesia Be a Classically Conditioned Response in Humans? A Systematic Review and Meta-Analysis. Pain Med. 2016 Jun;17(6):1094-111. doi: 10.1093/pm/pnv044. Epub 2015 Dec 14. PMID 26814278
- [Background] Madden VJ, Bellan V, Russek LN, Camfferman D, Vlaeyen JWS, Moseley GL. Pain by Association? Experimental Modulation of Human Pain Thresholds Using Classical Conditioning. J Pain. 2016 Oct;17(10):1105-1115. doi: 10.1016/j.jpain.2016.06.012. Epub 2016 Jul 22. PMID 27452948
- [Background] Van den Bergh O, Stegen K, Van de Woestijne KP. Learning to have psychosomatic complaints: conditioning of respiratory behavior and somatic complaints in psychosomatic patients. Psychosom Med. 1997 Jan-Feb;59(1):13-23. doi: 10.1097/00006842-199701000-00003. PMID 9021862
- [Background] Verrender A, Loughran SP, Anderson V, Hillert L, Rubin GJ, Oftedal G, Croft RJ. IEI-EMF provocation case studies: A novel approach to testing sensitive individuals. Bioelectromagnetics. 2018 Feb;39(2):132-143. doi: 10.1002/bem.22095. Epub 2017 Nov 10. PMID 29125197
- [Background] Wiech K. Deconstructing the sensation of pain: The influence of cognitive processes on pain perception. Science. 2016 Nov 4;354(6312):584-587. doi: 10.1126/science.aaf8934. PMID 27811269
- [Background] Larun L, Brurberg KG, Odgaard-Jensen J, Price JR. Exercise therapy for chronic fatigue syndrome. Cochrane Database Syst Rev. 2019 Oct 2;10(10):CD003200. doi: 10.1002/14651858.CD003200.pub8. PMID 31577366
- [Background] van Dessel N, den Boeft M, van der Wouden JC, Kleinstauber M, Leone SS, Terluin B, Numans ME, van der Horst HE, van Marwijk H. Non-pharmacological interventions for somatoform disorders and medically unexplained physical symptoms (MUPS) in adults. Cochrane Database Syst Rev. 2014 Nov 1;2014(11):CD011142. doi: 10.1002/14651858.CD011142.pub2. PMID 25362239
- [Background] Belleville S, Hudon C, Bier N, Brodeur C, Gilbert B, Grenier S, Ouellet MC, Viscogliosi C, Gauthier S. MEMO+: Efficacy, Durability and Effect of Cognitive Training and Psychosocial Intervention in Individuals with Mild Cognitive Impairment. J Am Geriatr Soc. 2018 Apr;66(4):655-663. doi: 10.1111/jgs.15192. Epub 2018 Jan 4. PMID 29313875
- [Background] Wenisch E, Cantegreil-Kallen I, De Rotrou J, Garrigue P, Moulin F, Batouche F, Richard A, De Sant'Anna M, Rigaud AS. Cognitive stimulation intervention for elders with mild cognitive impairment compared with normal aged subjects: preliminary results. Aging Clin Exp Res. 2007 Aug;19(4):316-22. doi: 10.1007/BF03324708. PMID 17726363
- [Background] Hallock H, Collins D, Lampit A, Deol K, Fleming J, Valenzuela M. Cognitive Training for Post-Acute Traumatic Brain Injury: A Systematic Review and Meta-Analysis. Front Hum Neurosci. 2016 Oct 27;10:537. doi: 10.3389/fnhum.2016.00537. eCollection 2016. PMID 27833541
- [Background] Mitolo M, Venneri A, Wilkinson ID, Sharrack B. Cognitive rehabilitation in multiple sclerosis: A systematic review. J Neurol Sci. 2015 Jul 15;354(1-2):1-9. doi: 10.1016/j.jns.2015.05.004. Epub 2015 May 9. PMID 25998261
- [Background] Ge S, Zhu Z, Wu B, McConnell ES. Technology-based cognitive training and rehabilitation interventions for individuals with mild cognitive impairment: a systematic review. BMC Geriatr. 2018 Sep 15;18(1):213. doi: 10.1186/s12877-018-0893-1. PMID 30219036
- [Background] Djabelkhir L, Wu YH, Vidal JS, Cristancho-Lacroix V, Marlats F, Lenoir H, Carno A, Rigaud AS. Computerized cognitive stimulation and engagement programs in older adults with mild cognitive impairment: comparing feasibility, acceptability, and cognitive and psychosocial effects. Clin Interv Aging. 2017 Nov 21;12:1967-1975. doi: 10.2147/CIA.S145769. eCollection 2017. PMID 29200836
- [Background] Pitron V. Vers un modèle cognitif bayésien du trouble à symptomatologie somatique [Thèse d'exercice]. [Paris]: Université Paris Descartes; 2017.
- [Background] Li J, Xia W, Zhan C, Liu S, Yin Z, Wang J, Chong Y, Zheng C, Fang X, Cheng W, Reinhardt JD. A telerehabilitation programme in post-discharge COVID-19 patients (TERECO): a randomised controlled trial. Thorax. 2022 Jul;77(7):697-706. doi: 10.1136/thoraxjnl-2021-217382. Epub 2021 Jul 26. PMID 34312316
- [Background] McNair, D. M., & Kahn, R. J. (1983). Self-assessment of cognitive deficits. Assessment in geriatric psychopharmacology, 137, 143.
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Van der Linden, M., Coyette, F., Poitrenaud, J., Kalafat, M., Calicis, F., Wyns, C., . . . Membres du GREMEM. (2004). L'épreuve de rappel libre/ rappel indicé à 16 items (RL/RI-16). In M. Van der Linden, S. Adam, A. Agniel, & Membres du GRENEM (Eds.), L'évaluation des troubles de la mémoire : présentation de quatre tests de mémoire épisodique avec leur étalonnage. (pp. 25-47). Marseille: Solal
- [Background] Tombaugh TN. Trail Making Test A and B: normative data stratified by age and education. Arch Clin Neuropsychol. 2004 Mar;19(2):203-14. doi: 10.1016/S0887-6177(03)00039-8. PMID 15010086
- [Background] Godefroy, O, et le GREFEX (Groupe de Réflexion pour l'Évaluation des Fonctions Exécutives) (2008). Fonctions exécutives et pathologies neurologiques et psychiatriques. Évaluation en pratique clinique. Marseille : Solal.
- [Background] Majerus, S. (2008). La mémoire verbale à court terme : un simple produit des interactions entre systèmes langagiers, attentionnels et de traitement de l'ordre sériel. Psychologie Française, 53, 327-341.
- [Background] Weschler, D. (2008). Weschler Adult Intelligence Scale (4th ed.). Peason.
- [Background] Cardebat D, Doyon B, Puel M, Goulet P, Joanette Y. [Formal and semantic lexical evocation in normal subjects. Performance and dynamics of production as a function of sex, age and educational level]. Acta Neurol Belg. 1990;90(4):207-17. French. PMID 2124031
- [Background] Giersky, F., & Ergis, AM. (2004). Les fluences verbales : aspects théoriques et nouvelles approches. Année Psychol, 104 : 331-360.
- [Background] Brickenkamp, R., Schmidt-Atzert, L., & Liepmann, D. (2015). d2-R: test d'attention concentrée révisé: manuel. Hogrefe.